CLINICAL TRIAL: NCT06225869
Title: Impact of Dopamine Replacement Therapy on Shame and Embarrassment-specific Processing and Its Clinical Relevance in Parkinson's Disease Patients
Brief Title: Effect of Dopamine on Specific Processing of Shame and Embarrassment in Parkinson's Disease
Acronym: BioDopa
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Vanessa Fleury, Principal Investigator, University Hospital, Geneva
Other Study IDs: 2022-00760
Record Dates: First submitted 2024-01-16; First posted 2024-01-26 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Assessments in ON and OFF levodopa state — Neurological assessment, neuropsychological assessment, and fMRI in ON and OFF levodopa state

SUMMARY:
Shame and embarrassment are two self-conscious emotions frequently experienced by Parkinson's disease (PD) patients. Shame and embarrassment scores strongly correlate with patient's quality of life, anxiety and depression ratings. However, the neurobiology of shame and embarrassment in PD and the influence of dopaminergic replacement therapy (DRT) is poorly understood.

The aim of this study is to characterize how brain structures and neuronal networks involved in Parkinson's disease-related shame, non-Parkinson's disease related shame and neutral control scenarios, are modulated by dopaminergic replacement therapy. For this purpose, functional MRI and connectivity measures between the basal ganglia and shame-related network will be analyzed while PD patients will perform a shame-induction task during both ON- (i.e. during the effect of DRT) and OFF-DRT (i.e. during the withdrawal of DRT) conditions. Correlation with clinical measures will be made.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease (PD) based on United Kingdom Parkinson's Disease Society Brain Bank Criteria
* Patients in the PD phase called "motor and non-motor fluctuations stage".
* Presence of motor and non-motor fluctuations are based on:

  1. For motor fluctuations: a score of 1 on item 4.1 and/or 1 on item 4.3 of the Movement Disorder Society Unified Parkinson's Disease Rating Scale IV
  2. For non-motor fluctuations: a score of 2 on item III of the Behavioral Assessment of Parkinson's Disease
* To be on dopaminergic replacement therapy.

Healthy controls:

subjects without any known central nervous system (CNS) lesion or CNS clinical signs on examination

Exclusion Criteria:

* Age greater than 80 years
* Dementia or mild cognitive impairment based on a score <26 on the MOCA
* Ongoing depression with suicidal ideation
* Any clinically meaningful non-stable renal, hepatic, cardiovascular, respiratory cerebrovascular disease or other serious progressive physical diseases
* Participating in a pharmacological study
* Any MRI contraindications
* Intolerable "OFF" states when the effects of the PD medication wear off (e.g., severe pain, anxiety, depression at the end of the dose or in the morning upon waking)
* Inability to provide informed consent (legal guardianship)
* Inability to speak or read French.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PD patients will be recruited from the outpatient movement disorder clinic of the Neurology Department at the Geneva University Hospital (HUG). Patients, who participated in previous studies and who are now followed up by private physicians, could also be contacted by trained members of the clinic/research staff to propose the study.
  Flyers with a brief explanation of the project could also be distributed to the physicians to invite patients to consider participating and reach out to a staff member for further information.
  Healthy controls will be recruited among the patients' spouses and through advertisement placed in the HUG and the University Medical Centre.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Difference in BOLD activity in ON versus OFF state | fMRI at rest and during a shame induction task, 1 hour in ON state and 1 hour in OFF state
  Difference in brain Blood Oxygenation Level Dependent (BOLD) activity between ON-levodopa versus OFF-levodopa patients, as well as age-matched healthy controls during the imaginary ideation of PD-shame related scenarios, non-PD shame related scenarios as well as neutral scenarios.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Fleury, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital, Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No